CLINICAL TRIAL: NCT06494943
Title: Neoadjuvant IBI110 and Sintilimab in Combination with Chemotherapy in Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)- a Phase Ib Clinical Trial
Brief Title: Induction IBI110 and Sintilimab with Chemotherapy in LA HNSCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Professor, M.D., Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Insight 3.0
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: Immune checkpoint inhibitor; Neoadjuvant chemotherapy; Induction chemotherapy; PD-1 inhibitor; LAG-3 inhibitor
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — sintilimab; Paclitaxel; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort B: IBI110 and sintilimab and TP regimen (Experimental): The first phase is the dose-escalation stage, where fixed doses of IBI110 and sintilimab will be administered, and the doses of paclitaxel and cisplatin will be escalated to determine the Recommended Dose for expansion stage. This phase is divided into three dose groups: paclitaxel 135 mg/m² on day 2 and cisplatin 20 mg/m² on days 2-4; paclitaxel 150 mg/m² on day 2 and cisplatin 20 mg/m² on days 2-4; paclitaxel 175 mg/m² on day 2 and cisplatin 25 mg/m² on days 2-4. The accelerated dose-escalation method will be used.
  The second phase is the fixed-dose expansion stage. They will receive the recommended doses of paclitaxel and cisplatin, combined with IBI110 200 mg on day 1 every 3 weeks administered intravenously, and sintilimab 200 mg on day 1 every 3 weeks administered intravenously.
  All subjects will undergo radical surgery after neoadjuvant therapy. Adjuvant radiotherapy (chemoradiotherapy) will be administered postoperatively based on pathological factors as appropriate.
  Interventions: Drug: Sintilimab; Drug: IBI110; Drug: Paclitaxel; Drug: Cis Platinum; Procedure: Surgery; Radiation: Adjuvant radiation
- Cohort A: sintilimab and TP regimen (Experimental): The enrolled patients will receive paclitaxel 175 mg/m² on day 2 and cisplatin 25 mg/m² on days 2-4, combined with sintilimab 200 mg on day 1 every 3 weeks administered intravenously, for a total of two cycles. All subjects will undergo radical surgery after neoadjuvant therapy. Adjuvant radiotherapy (chemoradiotherapy) will be administered postoperatively based on pathological factors as appropriate.

INTERVENTIONS:
Drug: Sintilimab — PD-1 inhibitor
  Arms: Cohort B: IBI110 and sintilimab and TP regimen
Drug: IBI110 — LAG-3 inhibitor
  Arms: Cohort B: IBI110 and sintilimab and TP regimen
Drug: Paclitaxel — Chemotherapy
  Arms: Cohort B: IBI110 and sintilimab and TP regimen
Drug: Cis Platinum — Chemotherapy
  Arms: Cohort B: IBI110 and sintilimab and TP regimen
Procedure: Surgery — Definitive surgery
  Arms: Cohort B: IBI110 and sintilimab and TP regimen
Radiation: Adjuvant radiation — Adjuvant radiotherapy or chemoradiotherapy based on post-operative pathologic findings.
  Arms: Cohort B: IBI110 and sintilimab and TP regimen

SUMMARY:
This study aims to investigate the efficacy and safety of combining sintilimab and the TP regimen with/without IBI110 for neoadjuvant chemotherapy in resectable locally advanced head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
The NCCN guidelines recommend that for resectable locally advanced HNSCC, the recommended treatment include surgery combined with postoperative adjuvant radiotherapy (chemoradiotherapy), or concurrent chemoradiotherapy; for locally extensive HNSCC, the guidelines recommend considering neoadjuvant chemotherapy, with subsequent selection of surgery or chemoradiotherapy based on the efficacy of the neoadjuvant chemotherapy. In recent years, multiple studies have shown that combining PD-1 inhibitors with neoadjuvant chemotherapy may help improve the pathological response rate of surgical resection.

LAG-3 (Lymphocyte Activation Gene 3) is a cell surface molecule co-expressed with CD4 and CD8 on activated CD4+ and CD8+ T cells, natural killer (NK) cells, B cells, and dendritic cells. LAG-3 is an activation-induced T cell receptor (TCR) co-receptor with high affinity for major histocompatibility complex (MHC) class II molecules, and it can directly inhibit TCR signal transduction in the immune response through its interaction with MHC II.

IBI110 can directly bind to LAG-3 on T cells, blocking the interaction between LAG-3 and MHC II, thereby relieving the inhibitory effect of LAG-3 on T cell activation and enhancing the anti-tumor immune response of T cells. Additionally, LAG-3 and PD-1 are both immune checkpoint receptors. Co-inhibition of LAG-3 and PD-1 can enhance immune responses and inhibit tumor growth. Therefore, IBI110 and its combination therapy with PD-1 monoclonal antibodies have great development potential in the treatment of locally advanced, recurrent, and late-stage solid tumors.

Based on the aforementioned foundation, this study intends to enroll patients with resectable locally advanced head and neck squamous cell carcinoma (HNSCC). The treatment protocol will involve neoadjuvant therapy and the TP regimen (paclitaxel and cisplatin), with/without IBI110 for neoadjuvant chemotherapy. Following neoadjuvant therapy, patients will undergo radical surgery, and adjuvant radiotherapy (chemoradiotherapy) will be administered postoperatively based on pathological risk factors as appropriate. The primary endpoints of the study are efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and willing to complete the study as per the protocol;
2. Age ≥ 18 years and ≤ 75 years;
3. Histologically confirmed head and neck squamous cell carcinoma, including primary sites in the oropharynx, oral cavity, larynx, and hypopharynx;
4. Resectable locally advanced head and neck squamous cell carcinoma (AJCC 8th edition: Stage III-IVB);
5. At least one measurable lesion before treatment, meeting the RECIST 1.1 criteria for "measurable disease";
6. Expected survival > 3 months;
7. ECOG performance status 0-1;
8. Adequate organ function meeting the following criteria:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   2. Platelet count ≥ 100 × 10^9/L;
   3. Hemoglobin ≥ 9 g/dL;
   4. Serum albumin ≥ 2.8 g/dL;
   5. Total bilirubin ≤ 1.5 × ULN, ALT, AST, and/or ALP ≤ 3 × ULN;
   6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 60 mL/min (Cockcroft-Gault, see Appendix III);
   7. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5 × ULN (Patients on stable doses of anticoagulants such as low-molecular-weight heparin or warfarin with INR within the therapeutic range may be screened);
9. Patients with HBV infection and inactive/asymptomatic HBV carriers, or those with chronic or active HBV, may be enrolled if HBV DNA < 500 IU/mL (or 2500 copies/mL) at screening. Patients with positive HCV antibodies may be enrolled if HCV-RNA is negative at screening;
10. Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days before treatment and use medically accepted contraception (e.g., intrauterine device, contraceptive pills, or condoms) during the study and for at least 3 months after the last dose of sintilimab and 6 months after the last dose of chemotherapy;
11. Non-sterilized male participants must agree to use medically accepted contraception (e.g., intrauterine device, contraceptive pills, or condoms) during the study and for at least 3 months after the last dose of toripalimab and 6 months after the last dose of chemotherapy.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. History of or concurrent other malignancies (excluding those that have been cured with a cancer-free survival period of more than 5 years, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma);
2. Receipt of any of the following treatments:

   1. Any investigational drug within 4 weeks prior to the first use of the study drug;
   2. Concurrent participation in another clinical study, unless it is an observational (non-interventional) clinical study;
   3. Systemic treatment with corticosteroids (daily dose >10 mg prednisone equivalent) or other immunosuppressive drugs within 2 weeks before the first use of the study drug, except for corticosteroids used for local inflammation and prevention of allergies, nausea, and vomiting. Special cases need to be discussed with the investigator. Inhaled or topical steroids and adrenal corticosteroid replacement therapy with doses >10 mg/day prednisone equivalent are allowed in the absence of active autoimmune disease;
   4. Anti-tumor vaccination or live vaccination within 4 weeks prior to the first administration of the study drug (for COVID-19 vaccination, the interval between vaccination and treatment should be more than 2 weeks);
   5. Major surgery or severe trauma within 4 weeks prior to the first use of the study drug;
3. Uncontrolled cardiac clinical symptoms or diseases, such as:

   1. Heart failure of NYHA class II or higher;
   2. Unstable angina;
   3. Myocardial infarction within 1 year;
   4. Clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
4. Severe infections (CTCAE > Grade 2) within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, or complications of infections. Baseline chest imaging indicating active pulmonary inflammation, symptoms and signs of infection within 4 weeks prior to the first use of the study drug, or requiring oral or intravenous antibiotics;
5. Active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); except for autoimmune-mediated hypothyroidism treated with a stable dose of thyroid replacement hormone, type 1 diabetes with a stable dose of insulin, vitiligo, or childhood asthma/allergies that have resolved without intervention in adulthood;
6. History of immunodeficiency, including positive HIV test, other acquired or congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation;
7. History of interstitial lung disease (excluding radiation pneumonitis that did not require steroid treatment) or non-infectious pneumonia;
8. Active pulmonary tuberculosis infection identified by history or CT scan, or a history of active pulmonary tuberculosis infection within 1 year prior to enrollment, or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal treatment;
9. Participants with active hepatitis B (HBV DNA ≥500 IU/mL or 2500 copies/mL) or hepatitis C (positive hepatitis C antibody and HCV-RNA above the lower limit of detection by the assay);
10. Known history of psychiatric drug abuse, alcoholism, or drug addiction;
11. Pregnant or breastfeeding women;
12. Other factors deemed by the investigator that could lead to forced early termination of the study, such as severe concomitant disease (including mental illness) requiring combined treatment, severely abnormal laboratory test values, or family or social factors that may affect the safety of the participant or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response | Up to 3 months, post-surgery
  The major pathological response rate (MPR rate), defined as the presence of residual tumor components ≤10% in tumor bed of the primary tumor site and cervical lymph node.
Adverse Events related to treatment | Up to 4 months
  Adverse Events related to treatment of sintilimab, IBI110, paclitaxel and cisplatin, per Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Pathologic complete response rate | Up to 3 months, post-surgery
  Pathologic complete response rate
Objective response rate | Up to 2 months, prior to surgery
  Objective response rate of primary tumor and metastatic lymph nodes, per RECIST 1.1 criteria
Progression-free survival rate | Up to 2 years
  Progression-free survival rate
Overall survival rate | Up to 2 years
  Overall survival rate
Quality of life asessment | Up to 2 months, prior to surgery
  Quality of life evaluation, based on EORTC QLQ-H&N35 criteria

OTHER OUTCOMES:
Tumor Mutation Burden | Up to 2 months, prior to surgery
  A measurement of mutations carried by tumor cells. It is a predictive biomarker being studied to evaluate its association with response to the study therapy, which may help to plan the best treatment. Tumors that have a high number of mutations appear to be more likely to respond to certain types of immunotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD sharing will be based on the decision of pricinpal investigator, after consultation of potential use of the data.

REFERENCES:
- [Background] Ou X, Zhai R, Wei W, Chen J, Ou D, Liao T, Xu T, Zhu Y, Wang Y, Huang S, Shi R, Wu B, Chen T, Li Y, Yang Z, Zhou C, Liu Y, Jiang Z, Zeng M, Liu X, Ji D, Ying H, Zhang Z, Hu C, Lu X, Ji Q, He X, Wang Y. Induction Toripalimab and Chemotherapy for Organ Preservation in Locally Advanced Laryngeal and Hypopharyngeal Cancer: A Single-Arm Phase II Clinical Trial. Clin Cancer Res. 2024 Jan 17;30(2):344-355. doi: 10.1158/1078-0432.CCR-23-2398. PMID 37955629
- [Background] Long L, Zhang X, Chen F, Pan Q, Phiphatwatchara P, Zeng Y, Chen H. The promising immune checkpoint LAG-3: from tumor microenvironment to cancer immunotherapy. Genes Cancer. 2018 May;9(5-6):176-189. doi: 10.18632/genesandcancer.180. PMID 30603054
- [Background] Tawbi HA, Schadendorf D, Lipson EJ, Ascierto PA, Matamala L, Castillo Gutierrez E, Rutkowski P, Gogas HJ, Lao CD, De Menezes JJ, Dalle S, Arance A, Grob JJ, Srivastava S, Abaskharoun M, Hamilton M, Keidel S, Simonsen KL, Sobiesk AM, Li B, Hodi FS, Long GV; RELATIVITY-047 Investigators. Relatlimab and Nivolumab versus Nivolumab in Untreated Advanced Melanoma. N Engl J Med. 2022 Jan 6;386(1):24-34. doi: 10.1056/NEJMoa2109970. PMID 34986285